CLINICAL TRIAL: NCT06802523
Title: A Phase I Study of Lintuzumab-Ac-225 in Combination With Venetoclax and ASTX-727 in Adults With Newly Diagnosed AML
Brief Title: Testing the Combination of Targeted Radiotherapy With Anti-Cancer Drugs, Venetoclax and ASTX-727, to Improve Outcomes for Adults With Newly Diagnosed Acute Myeloid Leukemia
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug Supply Issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-00575; NCI-2025-00575 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10653 (Other: Yale University Cancer Center LAO); 10653 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2025-01-29; First posted 2025-01-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Actinium; Specimen Handling; Biopsy; decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Schedule 1 (lintuzumab-Ac225, venetoclax, ASTX-727) (Experimental): INDUCTION: Patients receive lintuzumab-Ac225 IV over 30 minutes on day 8, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 1.
  RE-INDUCTION: Patients with CR,PR or NR after cycle 1 receive lintuzumab-Ac225 IV over 30 minutes on day 8, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 2.
  MAINTENANCE/CONSOLIDATION: Patients with CRi, CRh, or MLFS after cycle 1 receive venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Additionally, patients undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.
  Interventions: Radiation: Actinium Ac 225 Lintuzumab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- Schedule 2 (lintuzumab-Ac225, venetoclax, ASTX-727) (Experimental): INDUCTION: Patients receive lintuzumab-Ac225 V over 30 minutes on day 1, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 1.
  RE-INDUCTION: Patients with CR, PR or NR receive lintuzumab-Ac225 IV over 30 minutes on day 1, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 2.
  MAINTENANCE/CONSOLIDATION: Patients with CRi, CRh, or MLFS after cycle 1 receive venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Additionally, patients undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.
  Interventions: Radiation: Actinium Ac 225 Lintuzumab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax

INTERVENTIONS:
Radiation: Actinium Ac 225 Lintuzumab — Given IV
  Other Names: 225Ac-HuM195; Actimab-A; Actinium (225Ac) Lintuzumab Satetraxetan; Actinium-225-Labeled Humanized Anti-CD33 Monoclonal Antibody HuM195; LINTUZUMAB SATETRAXETAN AC-225; SGN-33 AC-225
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of lintuzumab-Ac225 in combination with venetoclax and ASTX-727, and how well they work in treating patients with newly diagnosed acute myeloid leukemia (AML). Lintuzumab-Ac225 is a monoclonal antibody, called lintuzumab, linked to a radioactive agent called actinium Ac 225. Lintuzumab attaches to CD33 positive cancer cells in a targeted way and delivers actinium Ac 225 to kill them. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. ASTX-727 is a combination of two drugs, cedazuridine and decitabine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Giving lintuzumab-Ac225 in combination with venetoclax and ASTX-727 may be safe and tolerable in treating patients with newly diagnosed AML and may improve the chance of going into remission and staying in remission for a longer period of time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine recommended phase 2 dose (RP2D) of actinium Ac 225 lintuzumab (lintuzumab-Ac225) when used in combination with venetoclax and decitabine and cedazuridine (ASTX-727).

SECONDARY OBJECTIVES:

I. To determine the maximum tolerated dose of lintuzumab-Ac225 when used in combination with venetoclax and ASTX-727.

II. To describe the frequency and severity of adverse events of patients treated on study, including cytopenia and organ toxicity after second dose of lintuzumab-Ac225.

III. To determine the rate and time to complete remission (CR), complete remission with incomplete hematologic recovery (Cri), and complete remission with partial hematologic recovery (CRh).

IV. To determine the rate and time to achieve CR/Cri/CRh without minimal residual disease (MRD) by multiparameter flow cytometry (MFC).

V. To determine the duration of remission, event-free and overall survival of patients.

VI. To evaluate and compare the clinical activity and toxicity between two lintuzumab-Ac225 administration schedules.

EXPLORATORY OBJECTIVES:

I. To correlate CD33 expression on AML cells with response to lintuzumab-Ac225 in combination with venetoclax and ASTX-727.

II. To evaluate CD33 isoforms as a variable for response to lintuzumab-Ac225 combination with venetoclax and ASTX-727.

OUTLINE: This is a dose-escalation study of lintuzumab-Ac225 in combination with venetoclax and ASTX-727. During dose-escalation phase, patients are randomized to 1 of 2 schedules.

SCHEDULE 1:

INDUCTION: Patients receive lintuzumab-Ac225 intravenously (IV) over 30 minutes on day 8, venetoclax orally (PO) once daily (QD) on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 1.

RE-INDUCTION: Patients with CR, partial response (PR) or no response (NR) after cycle 1 receive lintuzumab-Ac225 IV over 30 minutes on day 8, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 2.

MAINTENANCE/CONSOLIDATION: Patients with CRi, CRh, or morphologic leukemia-free state (MLFS) after cycle 1 receive venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.

SCHEDULE 2:

INDUCTION: Patients receive lintuzumab-Ac225 V over 30 minutes on day 1, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 1.

RE-INDUCTION: Patients with CR, PR or NR receive lintuzumab-Ac225 IV over 30 minutes on day 1, venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of cycle 2.

MAINTENANCE/CONSOLIDATION: Patients with CRi, CRh, or MLFS after cycle 1 receive venetoclax PO QD on days 1-28 and ASTX-727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of acute myeloid leukemia (AML) according to 2022 World Health Organization (WHO) criteria
* Evidence of CD33 expression in more than 25% of bone marrow blasts by flow cytometry determined by local assessment
* Patients must be considered ineligible for induction therapy defined by the following

  * ≥ 75 years of age; OR
  * <75 years of age with at least one of the following co-morbidities or high-risk genetic features. Geriatric assessment and other tools to assess frailty have not been validated in patients with AML, and therefore will not be used to assess eligibility

    * Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or 3;
    * Cardiac history of congestive heart failure (CHF) requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina;
    * Diffusion capacity of lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume in 1 second (FEV1) ≤ 65%;
    * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × upper limit of normal (ULN)
    * Patents with high risk genetic features based on local testing

      * inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2)
      * t(3q26.2;v)
      * -5 or del(5q); -7; -17/abnormal(17p)
      * Complex karyotype or monosomal karyotype as defined by ELN 2022
      * Mutated TP53
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of linituzumab-Ac-225 in combination with venetoclax and ASTX-727 in patients < 18 years of age, children are excluded from this study
* ECOG performance status 0-3 (Karnofsky ≥ 60%). For patients with ECOG performance status of 3, the decline in status should be due to AML per investigator's determination
* Total bilirubin ≤ 3.0x institutional ULN unless considered due to Gilbert syndrome
* Aspartate aminotransferase (AST)(serum gluatmic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* Creatinine clearance ≥ 60 ml/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification. Patients with heart failure must have NYHA functional class congestive heart failure (CHF) II or below to be eligible
* Hydroxyurea, cytarabine or leukopheresis are allowed for management of hyperleukocytosis, before initiation of study therapy. All-trans retinoic acid (ATRA) given emergently for suspected acute promyelocytic leukemia (APL) is also allowed. White blood cell (WBC) count must be < 25 x 10^9/L to start on study therapy per venetoclax label. Hydroxyurea and ATRA may be administered up to one day prior to start of study treatment
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Patients with favorable risk AML per the European LeukemiaNet (ELN) 2022 criteria
* Active central nervous system (CNS) involvement of AML requiring therapy
* Prior therapy with radiopharmaceuticals or external beam radiation therapy (EBRT)
* Previous therapy with venetoclax or other BCL-2 directed therapy
* Patients with Fridericia-corrected QT interval (QTcF) > 450ms at screening. QTcF will be calculated as the mean of the QTcF value from three separate electrocardiography (EKGs)
* Receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to venetoclax or ASTX-727
* Uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous per investigators opinion
* Pregnant women are excluded from this study because lintuzumab-Ac225 is a radiotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lintuzumab-Ac225, breastfeeding should be discontinued if the mother is treated with lintuzumab-Ac225. These potential risks may also apply to other agents used in this study

  * Women of child-bearing potential must agree to use adequate contraception (hormonal birth control or abstinence) prior to study entry and for the duration of study participation, and for 6 months following completion of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception (latex or synthetic condom or abstinence) prior to the study, for the duration of study participation, and 3 months after completion of the study
* Patients unable to swallow tablets/capsules and patients with malabsorption syndrome or other conditions that may interfere with the oral administration of medications are not eligible
* Patients who have had chemotherapy, targeted small molecule therapy (aside from imatinib, dasatinib, or nilotinib, hydroxyurea, cytarabine or ATRA),within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study are not eligible
* Prior allogenic stem cell transplant
* Patients who received a live vaccine within 30 days of planned start of study therapy

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist, registered trademark) are live attenuated vaccines, and are not allowed
* Patients who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit within 3 days prior to the initiation of study treatment and are unwilling to discontinue consumption of these throughout the receipt of study drugs
* Patients who are unable to take spironolactone or eplerenone due to intolerance, allergy, drug-drug interactions, or for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2026-04-21 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 28 days after the start of induction (up to 42 days for persistent neutropenia and thrombocytopenia)
  Adverse events (AEs) will be described and graded using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Overall response rate (ORR) | Up to 5 years
  Will include patients with complete remission (CR), complete remission with partial hematologic recovery (CRh), and complete remission with incomplete hematologic recovery (CRi). ORR and its 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Maximum tolerated dose of lintuzumab Ac-225 when used in combination with venetoclax and ASTX-727 | Up to completion of dose-escalation phase (Part A)
  Will be determined based on the totality of safety (specifically cytopenia), tolerability, clinical activity, as appropriate.
Frequency and severity of AEs | Up to 30 days after last dose of study treatment
  Will be assessed using CTCAE v 5.0. Toxicity by severity will be summarized using descriptive statistics. Will be listed for each dose level and the tabulations of AEs will also be produced by severity and by relationship to the study drug.
CR rate | Up to 5 years
  Will be evaluated per European Leukemia Network (ELN) 2022 response criteria. Will be defined as bone marrow blasts < 5%, absence of circulating blasts, absence of extramedullary disease, absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L (1,000uL), and platelet count ≥ 100 x 10^9/L (100 000/uL).
Time to CR | Up to 5 years
  Will be evaluated per ELN 2022 response criteria.
CRh rate | Up to 5 years
  Will be evaluated per ELN 2022 response criteria. Will be defined as ANC ≥ 0.5 x 10^9/L (500/uL) and platelet count ≥ 50 x 10^9/L (50 000/uL), otherwise all other CR criteria met.
Time to CRh | Up to 5 years
  Will be evaluated per ELN 2022 response criteria.
CRi rate | Up to 5 years
  Will be evaluated per ELN 2022 response criteria. All CR criteria except for residual neutropenia < 1.0 x 10^9/L (1,000/uL) or thrombocytopenia < 100 x 10^9/L (100 000/uL).
Time to CRi | Up to 5 years
  All CR criteria except for residual neutropenia < 1.0 × 109/L (1,000/µL) or thrombocytopenia < 100 × 109/L (100 000/µL)
CR rate without minimal residual disease (MRD) | At end of induction and end of first and third consolidation cycles (cycle length = 28 days), assessed up to 5 years
  Will be defined as CR with one or fewer residual leukemic blasts per 1,000 leukocytes as detected by multi-parameter flow cytometry (MFC). CR rate without MRD and its 95% confidence interval will be calculated.
CRh rate without MRD | At end of induction and end of first and third consolidation cycles (cycle length = 28 days), assessed up to 5 years
  Will be defined as CRh with one or fewer residual leukemic blasts per 1,000 leukocytes as detected by MFC. CRh rate without MRD and its 95% confidence interval will be calculated.
CRi rate without MRD | At end of induction and end of first and third consolidation cycles (cycle length = 28 days), assessed up to 5 years
  Will be defined as CRi with one or fewer residual leukemic blasts per 1,000 leukocytes as detected by MFC. CRi rate without MRD and its 95% confidence interval will be calculated.
Time to achieve CR without MRD | Up to 5 years
  Evaluated using MFC. CR without MRD and its 95% confidence interval will be calculated.
Time to achieve CRh without MRD | Up to 5 years
  Evaluated using MFC. CRh without MRD and its 95% confidence interval will be calculated.
Time to achieve CRi without MRD | Up to 5 years
  Evaluated using MFC. CRi without MRD and its 95% confidence interval will be calculated.
Duration of remission | From day of achieving CR, CRh, CRi to the date of hematological relapse or death from any cause, assessed up to 5 years
  Will be described using Kaplan-Meier product limit methods.
Progression free survival | Up to 5 years
  Will be described using Kaplan-Meier product limit methods.
Event-free survival | From day 1 of registration to the date of treatment failure, hematologic relapse from CR/CRh/CRi or death from any cause, whichever occurs first, assessed up to 5 years
  Will be described using Kaplan-Meier product limit methods.
Overall survival | From day 1 of registration to the date of death from any cause, assesesd up to 5 years
  Will be described using Kaplan-Meier product limit methods.
Clinical activity between two lintuzumab-Ac225 administration schedules | Up to 5 years
  Clinical activity will be defined as a patient achieving CR/CRi/CRh/morphologic leukemia-free state or partial response.
Toxicity between two lintuzumab-Ac225 administration schedules | Up to 5 years
  Will be assessed on the frequency or severity of AEs.

OTHER OUTCOMES:
Correlate CD33 expression on acute myeloid leukemia cells with response to lintuzumab-Ac225 in combination with venetoclax and ASTX-727 | Up to 5 years
  Will be assessed by flow cytometry and responses assessed by ELN 2022 response criteria. Will be summarized using descriptive statistics (means, median, and standard deviations) at each measurement time point and compared by paired t-test or Wilcoxon rank-sum test as appropriate.
CD33 isoforms as a variable for response to lintuzumab-Ac225 in combination with venetoclax and ASTX-727 | Up to 5 years
  Will be reported using Myeloseq-HD and responses will be assessed by ELN 2022 criteria. Will be summarized using descriptive statistics (means, median, and standard deviations) at each measurement time point and compared by paired t-test or Wilcoxon rank-sum test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Manu Pandey, Principal Investigator — Yale University Cancer Center LAO
Locations (1):
- Yale University Cancer Center LAO, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm